CLINICAL TRIAL: NCT02788331
Title: Revisiting the Volume-outcome Relationship in Surgery: Trends Analysis in French Hospitals
Brief Title: Trends in Volume-Outcome Relationship in Surgery
Acronym: TREVORS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0097
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Hospitals with increasing activity: Hospitals experiencing an increase in the volume of surgical procedures over the study period
  Interventions: Other: No intervention
- Hospitals with decreasing activity: Hospitals experiencing a decrease in the volume of surgical procedures over the study period
  Interventions: Other: No intervention
- Hospitals with stable activity: Hospitals experiencing no change in the volume of surgical procedures over the study period
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The explanatory mechanism of the relationship between the volume of surgical procedures performed by individual hospitals and the occurrence of serious adverse events is not clear. Based on the " practice makes perfect " dogma, we will explore whether a learning effect can explain the volume-outcome relationship for complex surgical procedures using a nationwide dataset. Especially, we assume that increasing volume of procedures over time may be associated with improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

All adults hospitalized to have one of the following major surgery: resection of oeso-gastric, intestinal and pancreatic cancer, treatment of intra-abdominal aortic aneurysm, coronary artery bypass graft, endarterectomy, hip fracture prosthesis

Exclusion Criteria:

* Hospitalization <24 hours
* Absence of surgical procedure
* Ambulatory care
* Palliative care
* Organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated in French public and private hospitals from January 2010 to December 2014
Sampling Method: Non-Probability Sample
Enrollment: 759518 (Actual)
Dates: Start 2016-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Inpatient mortality | Within 30 days of surgical procedure

SECONDARY OUTCOMES:
Reoperation occurence | Within 30 days of surgical procedure
Occurence of intensive or critical care unit stay | Within 30 days of surgical procedure
Occurence of postoperative complication | Within 30 days of surgical procedure
  Postoperative complication includes sepsis, pulmonary embolism or deep vein thrombosis and cardiac arrest
Occurence of unplanned hospital readmission | Within 30 days of hospital discharge related to index stay

CONTACTS AND LOCATIONS:
Overall Officials: Antoine DUCLOS, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Pôle Information Médicale Evaluation Recherche des Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Payet C, Polazzi S, Lifante JC, Cotte E, Grinberg D, Carty MJ, Sanchez S, Rabilloud M, Duclos A. Influence of trends in hospital volume over time on patient outcomes for high-risk surgery. BMC Health Serv Res. 2020 Apr 1;20(1):274. doi: 10.1186/s12913-020-05126-4. PMID 32238160